CLINICAL TRIAL: NCT01201980
Title: An Epidemiological Study to Evaluate Standard Daily Practice in Managing Patients With Arterial Hypertension and to Evaluate Patients' Quality of Life
Brief Title: An Epidemiological Study to Evaluate Standard Daily Practice in Managing Patients With Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRS-DUM-2010/2
Record Dates: First submitted 2010-09-14; First posted 2010-09-15 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension
Keywords: essential arterial hypertension; calcium antagonist
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subject population with essential arterial hypertension currently receiving treatment with a calcium antagonist

SUMMARY:
This study is aimed to evaluate response rate of the antihypertensive treatment with a calcium antagonist in real life practice, to evaluate patients' quality of life and to collect the following Serbia-specific epidemiology data on hypertension: demographic data, patents characteristics, and patients' management/treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject population with essential arterial hypertension currently receiving treatment with a calcium antagonist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Speciality care clinics
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
To evaluate proportion of patients on antihypertensive pharmacological treatment reaching SBP goals according to the ESC 2007 guidelines (<140 mmHg*). | 24 weeks

SECONDARY OUTCOMES:
To evaluate proportion of patients on antihypertensive pharmacological treatment reaching DBP goals according to the ESC 2007 guidelines (<90 mmHg*). | 24 weeks
To collect local epidemiological date on patients with hypertension (demographic data; hypertension management data: treatment, treatment changes and tolerability data). | 24 weeks
To evaluate patients quality of life after 12 and 24 weeks by using patients quality of life questionnaire | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: prof. dr Zorana Vasiljevic, Principal Investigator — Clinical Center of Serbia, Belgrade
Locations (8):
- Serbia (8):
  - Research Site, Belgrade
  - Research Site, Čačak
  - Research Site, Kamenitz
  - Research Site, Kragujevac
  - Research Site, Niš
  - Research Site, Niška Banja
  - Research Site, Pančevo
  - Research Site, Šabac